CLINICAL TRIAL: NCT06190197
Title: Prophylactic Antibiotics in Radical Cystectomy With Urinary Diversion
Brief Title: Prophylactic Antibiotics in Cystectomy With Diversion
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URO-2023-32133
Record Dates: First submitted 2023-12-13; First posted 2024-01-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Radical Cystectomy; Ileal Conduit; Neobladder Diversion

STUDY DESIGN:
Intervention Model Description: Randomized non-inferiority trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): No prophylactic antibiotics post operatively. Participants will receive antibiotics only if needed post-operatively such as for infection
- Treatment group (Experimental): Prophylactic antibiotics postoperatively.
  Interventions: Drug: Prophylactic antibiotics postoperatively.

INTERVENTIONS:
Drug: Prophylactic antibiotics postoperatively. — Prophylactic antibiotics postoperatively. All participants in this arm will receive nitrofurantoin 100 milligrams by mouth daily for either 10 or 21 days based on whether they had an ileal conduit or orthotopic neobladder, respectively, for the diversion. Participants will be instructed to swallow the capsule whole, preferably with food and at the same time each day. If a dose is forgotten, participants will be asked to take it when they remember and then take the next dose as usual. However, if they do not remember until the next dose, do not take extra capsules to make up the missed dose.
  Arms: Treatment group

SUMMARY:
Using a randomized 2 arm design, this study is being conducted to test for non-inferiority of no prophylactic antibiotic therapy versus the prophylactic oral antibiotic, nitrofurantoin, through comparison of rates of postoperative urinary tract infections within the 90-day postoperative period in patients with muscle invasive bladder cancer who undergo radical cystectomy with urinary diversion.

ELIGIBILITY:
Inclusion Criteria:

* Presence of muscle invasive bladder cancer and planning to undergo radical cystectomy with either ileal conduit or neobladder diversion.
* 18 years of age or older

Exclusion Criteria:

* Currently receiving antimicrobials for active infection
* Poor renal function with GFR < 30 ml/min
* Allergy to nitrofurantoin and unable to take an alternative antibiotic (cephalexin, trimethoprim-sulfamethoxazole, or ciprofloxacin)
* Pregnancy
* Unable to provide Informed consent
* Prior pelvic radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-13 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
test for non-inferiority | 90 days
  Test for non-inferiority of no antibiotic therapy versus the prophylactic oral antibiotic, nitrofurantoin, through comparison of rates of postoperative urinary tract infections within the 90-day postoperative period in patients with muscle invasive bladder cancer who undergo radical cystectomy with urinary diversion.
Difference in risk | 30 and 90 days
  Difference in risk of UTI within the first 30 days postoperative between treatment and no treatment groups.
  2-sample, 2-sided, t-test for a difference in proportions. Statistical hypothesis: H0: R1 - R2 = 0, Hα: R1 - R2 ≠ 0, where R1 is the risk (proportion) of UTI infection within the first 30 days, post operation, among those in the treatment group, and R2 among placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Hamed Ahmadi, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States